CLINICAL TRIAL: NCT00062127
Title: A Phase I Pharmacokinetic Interaction Study of Irinotecan (NSC616348) and Thalidomide (NSC66847) in Patients With Advanced Solid Tumors
Brief Title: Irinotecan and Thalidomide in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02537; 12044B; U01CA069852 (NIH); CDR0000304517 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Irinotecan; Thalidomide

ARMS (2):
- Arm I (irinotecan hydrochloride and thalidomide) (Experimental): Patients receive irinotecan IV over 90 minutes on days 1 and 22 and oral thalidomide once daily on days 15-28. All patients undergo disease re-evaluation at 6 weeks. Patients with stable or responsive disease may receive additional courses comprising irinotecan IV on day 1 and oral thalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: thalidomide; Other: pharmacological study
- Arm II (irinotecan hydrochloride and thalidomide) (Experimental): Patients receive irinotecan as in arm I and oral thalidomide once daily on days -6 to 7. All patients undergo disease re-evaluation at 6 weeks. Patients with stable or responsive disease may receive additional courses comprising irinotecan IV on day 1 and oral thalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: thalidomide; Other: pharmacological study

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy such as irinotecan use different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide with irinotecan may kill more tumor cells. This randomized phase I trial is studying the side effects and best way to give irinotecan and thalidomide in treating patients with metastatic or unresectable solid tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether thalidomide alters the pharmacokinetics of irinotecan in patients with advanced solid tumors.

II. Determine whether irinotecan alters the pharmacokinetics of thalidomide in these patients.

III. Determine the toxicity of this regimen in these patients. IV. Determine the observed antitumor response in patients treated with this regimen.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive irinotecan IV over 90 minutes on days 1 and 22 and oral thalidomide once daily on days 15-28.

Arm II: Patients receive irinotecan as in arm I and oral thalidomide once daily on days -6 to 7.

All patients undergo disease re-evaluation at 6 weeks. Patients with stable or responsive disease may receive additional courses comprising irinotecan IV on day 1 and oral thalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor

  * Metastatic or unresectable
  * Standard curative or palliative therapy is no longer effective or does not exist
* Measurable or assessable disease
* No uncontrolled brain metastases

  * Patients with brain metastases are eligible provided the following are true:

    * Stable neurologic status
    * At least 4 weeks since prior steroids or anticonvulsants
    * No neurologic dysfunction that would confound evaluation
* Performance status - Karnofsky 70-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of inflammatory bowel disease requiring therapy
* No chronic diarrhea syndromes
* No paralytic ileus
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use 2 forms of effective contraception, including 1 highly effective method, for at least 4 weeks before, during, and for 4 weeks after study participation
* Male patients must use effective barrier contraception during and for 4 weeks after study participation
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No uncontrolled seizure disorder
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection
* No significant traumatic injury within the past 28 days
* No serious, nonhealing wounds or ulcers
* No bone fractures
* No preexisting peripheral neuropathy grade 2 or greater
* At least 4 weeks since prior biologic therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* More than 28 days since prior major surgical procedure or open biopsy
* At least 4 weeks since prior investigational therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Effect of thalidomide on irinotecan hydrochloride pharmacokinetics | Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours
Effect of irinotecan hydrochloride on thalidomide pharmacokinetics | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 and 168 hours
Grade 3 or greater toxicities assessed using NCI CTC version 2.0 | Up to 3 years
  Will be summarized and analyzed using descriptive statistics. Exact 90% confidence intervals using the binomial distribution will be derived.
Response assessed using RECIST criteria | Up to 3 years
  Will be summarized and analyzed using descriptive statistics. Exact 90% confidence intervals using the binomial distribution will be derived.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States